CLINICAL TRIAL: NCT04410029
Title: Evaluation of a Decision Aid for Early Pregnancy Loss: a Pilot RCT Study
Brief Title: Evaluation of a Decision Aid for Early Pregnancy Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 842526
Record Dates: First submitted 2020-05-18; First posted 2020-06-01 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Early Pregnancy Loss
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Standard counseling + Healthwise Decision Aid
  Interventions: Other: Healthwise Decision Aid
- Control (Active Comparator): Standard counseling + a control informational handout.
  Interventions: Other: Control informational handout

INTERVENTIONS:
Other: Healthwise Decision Aid — Healthwise, a non-profit company that develops health content and patient information for hospitals, has created a decision aid for EPL management that is available through the EPIC Systems, an electronic medical record. Participants will be given this decision aid after EPL diagnosis and prior to options consultation with a provider.
  Arms: Intervention
Other: Control informational handout — Participants randomized to the control arm will be given an informational handout of treatment options after EPL diagnosis and prior to options consultation with a provider.
  Arms: Control

SUMMARY:
This study aims to determine the effect of the Healthwise decision aid on shared decision making in women undergoing management of early pregnancy loss.

DETAILED DESCRIPTION:
Early pregnancy loss (EPL) or miscarriage is a common problem occurring in 15-20% of pregnancies. EPL can safely be managed surgically, medically, or expectantly; patient preferences, together with provider recommendations, should be used to guide treatment decisions. The three management options differ substantially experientially for patients. Previous literature has shown that patients have preferences for treatment and higher satisfaction when treated according to their preferences. Decision aids provide individualized information to help patients clarify their priorities and personal values. There is good evidence that decision aids compared to usual care resulted in greater knowledge, more realistic expectations, lower decisional conflict relating to feeling informed, more active decision making, less people remaining undecided, and greater effect agreement on value and choice. Despite this, there is limited research on the extent of decisional conflict experienced by women undergoing treatment for EPL, or the effect of decision aids on decisional conflict. Furthermore, only a few decision aid tools are publicly available for this indication. The Healthwise decision aid tool receives high scores by the International Patient Decision Aid Standards Scale, and is readily available to patients within the clinical site's electronic medical record.

The investigators propose a pilot randomized control trial, enrolling 50 participants with EPL. The study will measure baseline decisional conflict, and randomize participants to counseling with or without the decision aid. The investigators intend to study the Decisional Conflict Scale at baseline and after counseling, knowledge scores, Decision Regret and the 9-item Shared Decision Making Questionnaire (SDM-Q9) after counseling. Study data can be used to inform future research and to identify patients with predictors for high decisional conflict. This study is the first step towards validation of a high-quality decision aid tool for patients undergoing EPL management. It will also be the first study to report on decisional conflict and regret in patients with early pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Definitive diagnosis of early intrauterine pregnancy loss (including anembryonic pregnancy and missed abortion [ultrasound examination demonstrates fetal pole without cardiac activity measuring between 5.3 and 7mm or an abnormal growth pattern diagnostic of EPL])
* 18 years or older
* Willing and able to give informed consent

Exclusion Criteria:

* Pregnancy of unknown anatomic location
* Unable to read English
* Prior options counseling with a Family Planning provider
* Clinically unstable requiring emergent surgical management with uterine evacuation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Decision Conflict Scale (DCS) | Post-counseling (one day)
  Low-literacy version of Decision Conflict Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No